CLINICAL TRIAL: NCT01117844
Title: Feasibility and Phase II Study Using Proton Radiation For WHO Grade I-III Meningiomas and Hemangiopericytomas
Brief Title: Proton Radiation For Meningiomas and Hemangiopericytomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 24309
Record Dates: First submitted 2010-04-28; First posted 2010-05-06 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Meningioma; Hemangiopericytoma
MeSH Terms: conditions — Meningioma; Hemangiopericytoma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton radiation (Experimental)
  Interventions: Radiation: Proton Radiation

INTERVENTIONS:
Radiation: Proton Radiation — Protons have been demonstrated for medulloblastoma and prostate cancer, and comparative treatment planning using protons versus photons have shown a clear advantage to protons in terms of dose distribution.

SUMMARY:
This is a Feasibility/Phase II study for patients with a diagnosis of WHO Grade I - III Meningioma & Hemangiopericytoma brain cancer to be given standard dose Proton radiotherapy. The study will be performed in two phases: first, feasibility with an enrollment of 12 patients and then Phase Page 8 of 20 II, with an enrollment of an additional 38 patients. All patients will also be given quality of life (QOL) instruments pretreatment, weekly during treatment, then q 3 months for year 1 post treatment, q6 months year 2 & 3 and yearly for year 4 & 5. Comparisons will be made between the enrolled subjects receiving proton therapy and the known literature on photon radiation. See section 2 for full objectives. The second phase will begin no earlier than 60 days after the last patient in the initial phase has completed treatment and once safety and feasibility has been verified. The secondary objectives will serve as the objectives for the second phase of the study.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objectives of this study are feasibility and safety. The study will be deemed infeasible if greater than 10% of pts experience one of the following:

* Patient cannot be given treatment because anatomy is such that a dosimetrically satisfactory treatment plan cannot be devised.

  (95% of target volume covered by 95% of the dose)
* Patient is unable to tolerate 20% of treatments (for any reason unable to set patient up within acceptable limits of tolerance, patient unable to tolerate treatment position or immobilization for duration of treatment) using proton radiotherapy (up to 80% of treatments could be delivered using photons).
* Patient is unable to complete all of his/her treatments within 7 days of estimated date of treatment completion or requires a treatment break greater than 5 days. Toxicity will be deemed unacceptable if greater than 20% of patients experience acute toxicity, as defined in Section 7.12.

Secondary Objectives:

* To assess acute side effects from irradiation using proton beam therapy in place of conventional photon beam therapy for the treatment of meningiomas.
* To assess quality of life outcomes, with a focus on the rate of severe fatigue at 6 and 12 months from end of treatment.
* To assess late complications from irradiation using proton beam therapy in place of conventional photon beam therapy for the treatment of meningiomas.
* To compare the dose distribution to tumor and surrounding normal structures using DVHs (Dose Volume Histograms) generated from the proton plan used to treat the patient and the photon plan generated for comparison purposes.
* To determine 1-yr local control and progression-free and overall survival using proton radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of WHO I-III meningiomas and hemangiopericytomas:

  1. WHO grade I :

     * Tumor that are newly diagnosed and tumors that are incompletely excised
     * Tumors that have recurred post resection
  2. WHO grade II:

     * Any tumor, either completely or incompletely excised
     * Any recurrent tumor
  3. WHO grade III and hemangiopericytoma:

     * Any tumor, either completely or incompletely excised
     * Any recurrent tumor
* Patients must have a Karnofsky Performance Status of 60. Age greater than 18 years Patients must be able to provide informed consent.
* Adequate bone marrow function: WBC greater than 4000/mm3, platelets greater than 100,000 mm3.
* Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms or other barrier methods etc.). Hysterectomy or menopause must be clinically documented.

Exclusion Criteria:

* Prior or simultaneous malignancies within the past two years (other than cutaneous squamous or basal cell carcinoma, melanoma in situ or thyroid carcinoma).
* Pregnant women, women planning to become pregnant and women that are nursing. Actively being treated on any other therapeutic research study.
* Prior radiation to the brain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-02-04 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and Safety | 90 days
  For proton to deemed feasible, no greater than 10% of patients should experience a) Patient cannot be given treatment because anatomy is such that a dosimetically satisfactory treatment plan cannot be devised, b) Patient is unable to tolerate 20% of treatments using proton therapy, and c) patient is unable to complete all treatments within 7 days of estimated date of treatment completion

SECONDARY OUTCOMES:
Late Toxicity | 90 days
  Late toxicity is defined as any grade 3 or higher toxicity, excluding seizures, observed later than 90 days from start of radiation therapy.
Fatigue - Brief Fatigue Inventory (BFI) | 5 Years
  Fatigue will be scored by the Brief Fatigue Inventory (BFI), a validated instrument, which will be evaluated at the following time points: Pre-radiation, weekly during treatment, at 3, 6, 9, 12 months post-radiation and then every 6 months. It is expected that BFI score will increase (as fatigue worsens) in the first 6-9 months post-radiation and then the BFI score will decrease (as fatigue improves) at 12-24 months post-radiation. Proton radiotherapy is expected to improve fatigue as compared to photon radiotherapy.
Health Related Quality of Life | 5 Years
  Health Related Quality of Life will be followed using the following: EQ-5D European Quality of Life Index, Fact-G Functional Assessment of Cancer Therapy-General (FACT-G), and Fact-BR Functional Assessment of Cancer Therapy-Brain. Fact-BR will be evaluated at the same time points as the BFI. EQ-5D and Fact-G will be evaluated at pre-radiation, at 3, 6, 9, 12 months postradiation and then every 6 months.
Cumulative total dose (Gy) to normal brain tissue | 8 Weeks
  Cumulative total dose (Gy) to normal brain tissue will be estimated based on dosimetry plans for both proton and photon. Proton radiotherapy is expected to decrease exposure to normal brain tissues.
Progression free survival (PFS) and overall survival (OS) | 5 Years
  PFS and OS are defined as the time from start of radiotherapy to first documented progression (event for PFS), death due to any cause or last patient contact alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the Unviersity of Pennsylvania, Philadelphia, Pennsylvania, United States